CLINICAL TRIAL: NCT04871789
Title: Optimization of Patients Long-term Management After the Coronavirus Infection COVID-19
Acronym: OPTIMIST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pirogov Russian National Research Medical University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID_2020_01
Record Dates: First submitted 2021-03-21; First posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with severe COVID-19 pneumonia
  Interventions: Diagnostic Test: Laboratory and instrumental examination
- Patients who had an asymptomatic COVID-19 3 months ago
  Interventions: Diagnostic Test: Laboratory and instrumental examination
- People who had close contact with patients with confirmed COVID-19 3 months ago but did not get sick
  Interventions: Diagnostic Test: Laboratory and instrumental examination

INTERVENTIONS:
Diagnostic Test: Laboratory and instrumental examination — All patients will undergo a comprehensive examination to identify the consequences of COVID-19

SUMMARY:
200 participants should be included in the study. There will be three groups: 100 participants with a severe course of the disease 3 months ago, 50 asymptomatic carriers of coronavirus infection 3 months ago and 50 people who were in close contact with patients with confirmed coronavirus infection 3 months ago, but not sick and without antibodies to SARS-CoV-2.

The study consists of two visits. At the first visit, after signing the consent to participate in the study, a screening examination will be performed to assess the criteria for inclusion and exclusion in the study.

At the second visit, patients who meet the inclusion criteria and do not have exclusion criteria will undergo clinical and instrumental examination, and biological samples will be collected for laboratory testing.

The aim of the study is to determine the most significant clinical and laboratory markers of the severity of the outcomes in the period of convalescence of the new coronavirus infection COVID-19. Clinical and laboratory indicators, the number and severity of signs of postcovid syndrome as well as pathological changes in lung tissue according to CT data in the group with covid pneumonia and indicators of immune status, hemostasis, endothelial dysfunction, inflammation, metabolism will be assessed.

ELIGIBILITY:
Inclusion Criteria:

For all groups:

* Informed consent signed by the patient.
* Men and women aged 18 and over.

Group COVID-19 (asymptomatic):

* Confirmed diagnosis of COVID-19 (positive SARS-CoV-2 RNA PCR test or history of IgM and / or IgG antibodies to SARS-CoV-2)
* Absence of any clinical symptoms associated with coronavirus infection.

Group Healthy:

* Contact with patients with symptomatic new coronavirus infection COVID-19 in the absence of personal protective equipment for at least 3 days.
* Absence of any clinical symptoms associated with coronavirus infection

Group COVID symptomatic:

* Confirmed diagnosis of previous COVID-19 (positive SARS-CoV-2 RNA PCR test or presence of IgM antibodies to SARS-CoV-2) in history.
* A severe course of COVID-19, characterized by one or more of the following symptoms:

  * Respiratory rate ≥ 30 in 1 min
  * Blood oxygen saturation (SpO2) ≤ 93%
  * The ratio of the partial tension of oxygen in arterial blood to the fraction of oxygen during inspiration (PaO2 / FiO2) <300
  * Lung tissue lesion> 50% and / or according to computed tomography CT-2 and higher
  * Septic shock / sepsis
  * Development of multiple organ failure
  * Cytokine storm

Exclusion Criteria:

* Pregnancy
* Covid-19 vaccination
* Any serious medical illness before coronavirus infection, as well as a permanent form of atrial fibrillation
* Regular intake of anti-inflammatory, antibacterial, cytostatic and immunosuppressive drugs
* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women aged 18 and over with asymptomatic or severe course of the novel coronavirus infection COVID-19, or who have been in close contact with patients with confirmed coronavirus infection, but who are not sick and do not have antibodies to SARS-CoV-2
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-05-15 (Estimated); Study Completion 2021-06-15 (Estimated)

PRIMARY OUTCOMES:
The presense of postcovid syndrome | through study completion, an average of 3 months
  Clinical and laboratory indicators The number and severity of signs of postcovid syndrome

SECONDARY OUTCOMES:
Pathological changes in lung tissue according to CT data | through study completion, an average of 3 months
  CT scan

CONTACTS AND LOCATIONS:
Locations (1):
- Russian Clinical Research Center for Gerontology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided